CLINICAL TRIAL: NCT01131637
Title: A Phase III, Multi-center,Randomized, Double-blind, Based on Standard Therapy, Placebo-controlled Study of the Survival of Recombinant Human Neuregulin-1β in Patients With Chronic Systolic Heart Failure
Brief Title: Study of the Survival of Recombinant Human Neuregulin-1β in Chronic Heart Failure (CHF) Patients
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor has designed another study to replace the current study
Sponsor: Zensun Sci. & Tech. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZS-01-301
Record Dates: First submitted 2010-05-25; First posted 2010-05-27 (Estimated); Last update posted 2017-12-21 (Actual); Status verified 2012-07

CONDITIONS: Chronic Heart Failure
Keywords: chronic heart failure; rhNRG-1; mortality

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rhNRG-1 (Experimental): recombinant human neuregulin-1
  Interventions: Drug: rhNRG-1
- placebo (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: rhNRG-1 — day1~day10:0.6ug/kg/day,10hours per day for vein infusion; week3~week25:0.8ug/kg/day,10minutes per time per week for vein injection
  Arms: rhNRG-1
Drug: placebo — day1~day10:0.6ug/kg/day,10hours per day for vein infusion; week3~week25:0.8ug/kg/day,10minutes per time per week for vein injection
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate efficacy of rhNRG-1 in reducing the death rate of heart failure.

DETAILED DESCRIPTION:
The mortality of chronic heart failure patients remains high, in spite of recent treatment. RhNRG-1(recombinant human neuregulin-1)directly work on the cardiomyocyte and restored the normal structure and function of it. Both the preclinical trial and phase II clinical trail have confirmed that rhNRG-1 effectively enhance the heart function and reverse the remodeling of left ventricular in heart failure animals and humans. In this study, we will evaluate efficacy of rhNRG-1 in reducing the death rate of heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 80, both sex.
2. Left ventricular ejection fraction (LVEF)≤40% (ECHO).
3. NYNA functional class III~Ⅳ.
4. Clinical symptom is steadily in the latest 1 week (no fluid retension, no weight gain).
5. Capable of signing the informed consent form.

Exclusion Criteria:

1. Patients with acute pulmonary edema or acute hemodynamic disorder.
2. Patients with right heart failure caused by pulmonary disease.
3. Patients diagnosed with pericardial effusion or pleural effusion.
4. Patients with myocardial infarction during the preceding 3 months.
5. Patients with constrictive pericarditis, significant valvular pathological change or congenital heart diseases, severe pulmonary artery hypertension.
6. Unstable angina pectoris.
7. Cardiac surgery or cerebrovascular accident within recent six months.
8. Preparing for heart transplantation.
9. Serious ventricular arrhythmia (multi-morphological premature ventricular contraction, frequent paroxysmal ventricular tachycardia).
10. Serious hepatic or renal dysfunction caused by organic pathological changes (Cr>3.0mg/dl, AST or ALT 10 times above the normal upper limit).
11. Serum potassium <3.2 mmol/L or >5.5 mmol/L.
12. Systolic blood pressure <90mmHg or >160mmHg.
13. Pregnant or plan to pregnant.
14. Patients who participated in any clinical trial in the recent three months.
15. Subject with a life expectancy less than 3 months as assessed by the investigator.
16. Serious nervous system diseases (Alzheimer's disease, advanced Parkinsonism).
17. History of any malignancy or suffering from cancer,or biopsy proven pre-malignant condition (eg DICS or cervical atypia).
18. Evidence (physical examination,CXR,ECHO or other tests) shows some active malignancy or adenoidal hypertrophy or neoplasm has effect on heart function or endocrine system, eg pheochromocytoma or hyperthyroidism.
19. Judging by the investigator, the patients could not complete the study or adhere to the study requirements (due to the management reasons or others).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 331 (Actual)
Dates: Start 2010-04; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
all cause mortality | one year

CONTACTS AND LOCATIONS:
Overall Officials: Runlin Gao, MD,Ph.D, Principal Investigator — Cardiovascular Institute and Fuwai Hospital
Locations (43):
- China (43):
  - General Hospital of Chinese People's Liberation Army, Beijing, Beijing Municipality
  - The First Hospital affiliated to Lanzhou University, Lanzhou, Gansu
  - Haikou Municipal Peoples Hospital, Haikou, Hainan
  - Bethune International Peace Hospital, Shijiazhuang, Hebei
  - Teda International Cardiovascular Hospital, Tianjin, Hebei
  - Daqing Oilfield General Hospital, Daqing, Heilongjiang
  - The First Hospital of Harbin Medical University, Haerbin, Heilongjiang
  - The First hospital affiliated to Zhengzhou University, Zhengzhou, Henan
  - Zhongnan Hospital of Wuhan University, Wuchang, Hubei
  - Tongji Hospital Affiliated to Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Provincial People's Hospital, Changsha, Hunan
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Jiangyin People's Hospital, Jiangyin, Jiangsu
  - Nanjing Drum Tower Hospital, Nanjing, Jiangsu
  - Zhongda Hospital, Southeast University, Nanjing, Jiangsu
  - The Second Hospital affiliated to Suzhou University, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical School, Xuzhou, Jiangsu
  - North Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The Affiliate Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The Second Hospital affiliated to Jilin University, Changchun, Jilin
  - The First Hospital affiliated to Dalian Medical University, Dalian, Liaoning
  - The first affiliated hospital of Liaoning medical college, Jinzhou, Liaoning
  - Liaoning Provincial People's Hospital, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - The First Hospital of China Medical Hospital, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - The Second Hospital of Shandong University, Jinan, Shandong
  - Shanxi Provincial People's Hospital, Xi’an, Shanxi
  - The second hospital of Xi'an jiaotong university, Xi’an, Shanxi
  - Huaxi Hospital of Sichuan University, Chengdu, Sichuan
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - The Xinqiao Hospital of Third Military Medical University, Chongqin, Sichuan
  - Kunming General Hospital of Chengdu Military Region, Kunming, Yunnan
  - The Second hospital affiliated to Kunming Medical and Pharmaceutical College, Kunming, Yunnan
  - Sir Run Run Shaw Hospital affiliated to School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - The First Hospital affiliated to School of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Beijing Anzhen Hospital, Affiliate of Capital University of Medical Sciences, Beijing
  - Beijing Chao Yang Hospital, Affiliate of Capital University of Medical Sciences, Beijing
  - Cardiovascular Institute and Fuwai Hospital, Beijing
  - Huashan Hospital affiliated to Fudan University, Shanghai
  - Renji Hospital, Medical School of Shanghai Jiaotong University, Shanghai
  - The first people's hospitial of Shanghai, Shanghai
  - The Sixth People's Hospital, Shanghai Jiaotong University, Shanghai